CLINICAL TRIAL: NCT01072955
Title: Efficacy And Safety Of Heparin In Patients With Cardiovascular Surgery Using Cardiopulmonary Bypass
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azidus Brasil (Industry)
Responsible Party: Dr. Alexandre Frederico, LAL Clinica
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HEPSBCCV1109BOV_EUR; version 2
Record Dates: First submitted 2010-02-19; First posted 2010-02-22 (Estimated); Last update posted 2011-01-28 (Estimated); Status verified 2011-01

CONDITIONS: Prevention of Venous Thromboembolism
MeSH Terms: interventions — Heparin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- heparin of bovine origin (Experimental): 5.000UI/mL bottle with 5mL
  Interventions: Biological: Bovine Heparin
- heparin of porcine origin (Active Comparator): 5000 USP Heparin Units / mL vial with 10 mL vial
  Interventions: Biological: Porcine heparin

INTERVENTIONS:
Biological: Bovine Heparin — 5.000UI/mL bottle with 5mL
  Arms: heparin of bovine origin
Biological: Porcine heparin — 5000 USP Heparin Units / mL vial with 10 mL vial
  Arms: heparin of porcine origin

SUMMARY:
The primary objective of this study is to verify, through a randomized, blinded, parallel clinical trial, the efficacy of bovine heparin from Eurofarma Laboratory product when compared to porcine heparin APP Pharmaceutical in patients undergoing surgery cardiovascular disease and who require cardiopulmonary bypass, through the control of hemostasis during and after surgery, based on measurements of markers of coagulation ACT, aPTT, anti-Xa heparin levels and the excessive blood loss (hemorrhage) after the end of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients who agree with all aspects of the study and sign the FICT;
* Patients of both sexes;
* Patients over the age of 18 years;
* Patients with indication for cardiac surgery requiring cardiopulmonary bypass.

Exclusion Criteria:

* Patients with hematological disorders that compromise the surgical outcome (eg, myeloproliferative disorders, anemia, Hb <11.0 g / dL, platelets <100,000 mm3);
* Patients with disorders of hemostasis (INR> 1.40) (APTTr> 1.40);
* Patients with renal impairment (creatinine> 1.50);
* Patients with deep hyperthermia;
* Liver disease (AST and ALT> 2 times that of the reference value);
* Patients with a history of allergy to heparin or protamine;
* Patients with a history of heparin-induced thrombocytopenia;
* infection (eg endocarditis, septicemia and pneumonia);
* Reoperations;
* Use of antiplatelet agents (clopidogrel and ticlopidine) for less than 7 days;
* Use of aspirin for less than 5 days;
* Use of heparin, low molecular weight less than 24 hours;
* Use of unfractionated heparin for less than 12 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2010-04; Primary Completion 2010-08 (Estimated); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
Coagulometric parameters markers heparin activity: ACT, APTT and Anti - Xa | (T0) Pre heparintion; (T1) Top of extracorporeal; (T2) Intraoperative period; (T3) End bypass; (T4) Postoperative

SECONDARY OUTCOMES:
Value of the total dose of heparin used, the activity and adequate reversal with the use of protamine. | (T0) Pre heparintion; (T1) Top of extracorporeal; (T2) Intraoperative period; (T3) End bypass; (T4) Postoperative

CONTACTS AND LOCATIONS:
Locations (1):
- LAL Clinica Pesquisa e Desenvolvimento Ltda, Valinhos, São Paulo, Brazil